CLINICAL TRIAL: NCT00840307
Title: Changes in Ectopic Fat Following Surgically Induced Weight Loss: Does it Explain the Resolution of Diabetes?
Brief Title: Changes in Ectopic Fat Following Surgically Induced Weight Loss
Status: Completed | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ildiko Lingvay, MD, MPH, MSCS, University of Texas Southwestern Medical Center
Other Study IDs: 072008-039; NIH Grant: 1K23RR024470-01
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Results first posted 2017-11-20 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Obesity; Type 2 Diabetes
Keywords: Obesity; Type 2 Diabetes; Gastric Banding
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study evaluates how ectopic fat (in the pancreas, heart, liver and skeletal muscle), visceral fat, and subcutaneous fat changes following surgically induced weight loss using gastric banding. The investigators also evaluate whether changes in pancreatic fat content correlate with improvement in beta-cell function.

DETAILED DESCRIPTION:
We are looking for volunteers for this study,wich involves 7 visits over a period of 13 months, the first visit taking place about 2 weeks prior to the planned surgery.

Visit 1 - baseline, before starting your pre-operative diet Visit 2 - just before the surgery Visit 3 - around the time your first band inflation occurs Visit 4 - 1 month after the band inflation Visit 5 - 3 months after the first band inflation Visit 6 - 6 months after the first band inflation Visit 7 - 12 months after the first band inflation

At each visit we do the following tests:

1. MRS to measure your fat in the liver, pancreas, heart, muscle (leg), subcutaneous fat and visceral fat.
2. Frequently sampled intravenous glucose tolerance test - it is a 3.5 hrs test which determines the amount of insulin your body produces and how well your own insulin is being used by the body
3. Body measurements (waist, hip circumference), cholesterol panel, liver function tests, HbA1c (to monitor diabetes control), blood pressure, weight.

We also do an oral glucose tolerance test to check for diabetes on 3 occasions: visit 1, visit 5 and at the end, visit 7.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years old
* Fully understanding and willing to undergo study procedures
* Available for follow-up
* Understand and willing to sign informed consent
* Pharmacologic agents with the potential to change ectopic fat content (i.e. pioglitazone) are allowed if the patient has been on a stable dose for at least 3 months and plans to continue the same dose for the duration of the study

Exclusion Criteria:

* Contraindication to MRI (i.e. metallic implants, severe claustrophobia, weight above 320lb)
* Contraindication to phlebotomy (i.e. no accessible veins, hemoglobin <10 mg/dL)
* History of pancreatic disease other than diabetes
* Regular use of more than 2 alcoholic drinks per day
* Pregnancy
* Non-English speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients already scheduled to undergo gastric banding within 1-2 months.
  This study does NOT pay for the bariatric surgery, eligible participants must already be scheduled to have the surgery performed by their own physician
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2008-08; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ildiko Lingvay, MD, MPH, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient With Gastric Band: 20 patients recruited from bariatric surgery clinic followed-up before surgery and for 12 months after inflation of the gastric band.
Period: Overall Study
Arm/Group | Patient With Gastric Band
Started | 20
Completed | 16
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | Patient With Gastric Band
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Pancreatic and Liver Triglyceride (Fat) Content
Description: Pancreatic triglyceride (fat) content measured by the magnetic resonance spectroscopy (MRS) technique in volunteers with a wide range of body mass index (BMI).
Time Frame: months after the first band inflation
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | Patient With Gastric Band
Number analyzed (Participants) | 16
percent
  Pancreatic fat | 6.44 [1.75 to 25.02]
  Liver fat | 2.08 [1.43 to 3.63]

ADVERSE EVENTS:
Time Frame: 13 months
Arm/Group | Patient With Gastric Band
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No